CLINICAL TRIAL: NCT04255888
Title: Clinical Evaluation of the Impact of Periodontal Phenotype on the Outcome of Laterally Positioned Flap in Isolated Gingival Recession
Brief Title: Periodontal Phenotype and Laterally Positioned Flap in Isolated Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anjali perio
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thick periodontal phenotype (Active Comparator): Laterally positioned flap will be performed in isolated gingival recession belonging thick periodontal phenotype .
  Interventions: Procedure: Laterally positioned flap in thick periodontal phenotype.
- Thin periodontal phenotype (Active Comparator): Laterally positioned flap will be performed in isolated gingival recession belonging thin periodontal phenotype .
  Interventions: Procedure: Laterally positioned flap in thin periodontal phenotype.

INTERVENTIONS:
Procedure: Laterally positioned flap in thick periodontal phenotype. — Laterally positioned flap will be performed in isolated gingival recession belonging thick periodontal phenotype .
  Arms: Thick periodontal phenotype
Procedure: Laterally positioned flap in thin periodontal phenotype. — Laterally positioned flap will be performed in isolated gingival recession belonging thin periodontal phenotype .
  Arms: Thin periodontal phenotype

SUMMARY:
The aim of this study is to estimate the effect of periodontal phenotype on the outcome of isolated gingival recession by laterally positioned flap.The primary objective of study is to assess the changes in gingival margin in the donor tooth after laterally positioned flap over a period of 6 months and to assess the influence of periodontal phenotype on the stability of results of root coverage achieved through laterally positioned flap. The secondary objective of this study is to evaluate root coverage by laterally positioned flap in thick periodontal phenotype and to evaluate root coverage by laterally positioned flap in thin periodontal phenotype.

DETAILED DESCRIPTION:
A variety of surgical techniques have been proposed to achieve successful and predictable root coverage. These include coronally advanced flap, lateral positioned flap (LPF) free gingival graft, free connective tissue graft, and guided tissue regeneration. LPF, originally described by Grupe and Warren in 1964 is one of the most commonly performed root coverage technique.The procedure has undergone various modification over the years .Staffileno and pfeifer and Heller advocated the use of split-thickness flap to minimize the potential risk for the development of recession in the donor tooth.Wood et al used re-entry procedures to compare crestal radicular bone responses to full and partial thickness flaps. They concluded that regardless of the flap procedure, loss of crestal bone depended on the periodontal phenotype.The term periodontal phenotype refers to phenotypic characteristic of bone and soft tissue that make up the periodontium. Periodontal phenotype is typically used to describe the buccolingual tissue thickness and gingival morphology. It is divided into thick flat and thin scalloped type. However there is a paucity of studies in the literature studying the effect periodontal phenotype on the root coverage obtained and its stability over time after LPF. Furthermore the impact of periodontal phenotype on the donor area in this procedure has not been explored. Therefore the present study is designed with the aim to evaluate the influence of periodontal phenotype on the outcome of root coverage by LPF.

ELIGIBILITY:
INCLUSION CRITERIA

* Isolated Miller's class I, class II, and class III gingival recession in the anterior region
* Gingival Recession depth should be ≥2mm.
* Width of keratinized gingiva ≥3 mm on the immediately adjacent tooth

EXCLUSION CRITERIA

* Patients with a history of systemic condition that might alter the course of disease and /or wound healing such as diabetes mellitus, immunologic disorders.
* Pregnant and lactating women .
* Non vital tooth
* Smokers
* Caries, cervical abrasion or restoration on the labial aspect of tooth with gingival recession.
* Periodontal surgical treatment during previous 24 months on the involved sites.
* Miller's class IV. All potential participants would be explained the need and design of study .Only those subjects who consented for the study will be included after obtaining an informed consent.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Root coverage | 6 months
  Root coverage as seen by Reduction in gingival recession depth and width

SECONDARY OUTCOMES:
Location of gingival margin and periodontal status in the donor site area | 6 months
  Distance from customised fabricated stent to gingival margin of donor and treated tooth

CONTACTS AND LOCATIONS:
Overall Officials: Anjali kothari, Principal Investigator — post graduate institute of dental sciences,rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
STUDY PROTOCOL
Supporting Information: Study Protocol